CLINICAL TRIAL: NCT02846480
Title: Benefits of Peri-surgical Physical Therapy in the Management of III and IV Grades of Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BEATRIZ SANCHEZ SANCHEZ (Other)
Collaborators: Hospital Universitario Principe de Asturias (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, BEATRIZ SANCHEZ SANCHEZ, PHD, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UAlcala_POP
Record Dates: First submitted 2016-07-15; First posted 2016-07-27 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2016-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Physical Therapy Modalities; Surgical Procedures, Operative; Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgical treatment+behavior therapy+physical therapy (Experimental): Including POP surgical treatment, and pre- post physical therapy to aim the posture, PFM awareness and the strengthening. They will be also informed and instructed on hygienic and behavioral education to prevent POP and urinary incontinence (behavior therapy).
  Interventions: Other: physical therapy; Other: surgical treatment; Other: behavior therapy
- surgical treatment+behavior therapy (Experimental): Including POP surgical treatment, and information and instruction about hygienic and behavioral education to prevent POP and urinary incontinence (behavior therapy).
  Interventions: Other: surgical treatment; Other: behavior therapy

INTERVENTIONS:
Other: physical therapy — Pre-surgical Physical Therapy: physical therapy aimed to correct the posture, to the awareness and the strengthening of the pelvic floor muscles.
  Post-surgical Physical Therapy: checking the correct contraction of the pelvic floor muscles and hypopressive exercises.
  Arms: surgical treatment+behavior therapy+physical therapy
Other: surgical treatment — Surgical correction of POP.
Other: behavior therapy — At hospital discharge, patients will receive a fact sheet on the sanitary and behavioral measures recommended for the prevention of POP and urinary incontinence (proper weight, prevent constipation, avoid weight bearing and cough and high impact exercise).

SUMMARY:
To find out the effectiveness of physical therapy associated with the surgical treatment over the simptoms and quality of life in III and IV grades of pelvic organ prolapse, patients will be randomly assigned to one of these groups: experimental group: pre-surgical and post-surgical physical therapy + behavioral education + surgical therapy. Control group: surgical treatment + behavioral education.

In both groups several physical therapy assessments will be undertaken: 1st before surgery; 2nd immediately after surgery; and after 6 weeks, 3th, 6th, 12th and 24th months post-surgery.

DETAILED DESCRIPTION:
Intervention in the experimental group, patients assigned to this group will receive:

* Pre-surgical physical therapy: 9 sessions of physical therapy aimed at correcting posture, to the awareness and the strengthening of the pelvic floor muscles. They will be also informed and instructed on hygienic and behavioral education to prevent pelvic organ prolapse and urinary incontinence. Each session will be about 45 minutes and 3 sessions will be held a week for 3 weeks.
* Post-surgical Physical Therapy:

  2. Hospital discharge patients will receive the same fact sheet on sanitary and behavioral measures recommended for the prevention of pelvic organ prolapse and urinary incontinence.

  3. 6th weeks after surgery: 8 physical therapy sessions (2 per week for 4 weeks) about 30 minutes to review hypopressive exercises and contractions of the pelvic floor.

Intervention in the control group, patients assigned to this group will receive:

After surgical correction of pelvic organ prolapse, at hospital discharge, patients will receive a fact sheet on the sanitary and behavioral measures recommended for the prevention of pelvic organ prolapse and urinary incontinence (proper weight, prevent constipation, avoid weight bearing and cough and high impact exercise). No physical therapy intervention will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive women diagnosed with grade III and IV pelvic organ prolapse, which would be operated for this reason at the Asturias Prince Hospital (Madrid-Spain).

Exclusion Criteria:

* Women diagnosed with different III / IV grade of POP or a history of conservative treatment not from the subproject "Physiotherapy in the POP grades I and II", or a history of POP surgery, or concurrent conditions that would be affect the treatment (neurological, gynecological or urological), or recurrent urinary infection or hematuria, or those III / IV grades in POP which is contraindicated or not possible to perform surgery.
* Pregnant women or women with a vaginal birth in the last six months.
* Women with cognitive limitations to understand the information, answer questionnaires, consent and / or participate in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The SF-12 Health Survey (SF-12) Spanish version | up to 24th months post-surgery.
Assessment of pelvic floor muscles strength with Modified Oxford Scale and vaginal perineometry, vaginal dynamometry | up to 24th months post-surgery.
International Consultation on Incontinences Short Form (ICIQ-SF) Spanish version. | up to 24th months post-surgery.

SECONDARY OUTCOMES:
Urinary symptoms (urinary frequency, nocturia, urgency, incontinence, coital incontinence, nocturnal enuresis, frequency of urinary tract infections, dysuria and urinary difficulty). | up to 24th months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Maria José Yuste, PHD, Study Director — Alcalá University; María Torres, PHD, Study Chair — Alcalá University; Beatriz Navarro, PHD, Study Chair — Alcalá University

IPD SHARING:
Plan to Share IPD: No